CLINICAL TRIAL: NCT02051751
Title: A Phase Ib Open Label Dose Finding Study of BYL719 in Combination With Paclitaxel in Advanced Solid Tumors Followed by Two Expansion Phases in Locally Advanced/Metastatic Chemotherapy Naive HER2 Negative Breast Cancer Patients (HER2- mBC) and in Recurrent and Metastatic Head-and-neck Squamous Cell Carcinoma Patients (HNSCC) Pre-treated With Platinum Based Therapy
Brief Title: A Study to Evaluate the Potential Benefit of the Addition of BYL719 to Paclitaxel in the Treatment of Breast Cancer and Head-and-neck Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CBYL719Z2101
Record Dates: First submitted 2014-01-21; First posted 2014-01-31 (Estimated); Last update posted 2020-12-08 (Actual); Status verified 2020-12

CONDITIONS: Neoplasms, Breast Neoplasms, Head and Neck Neoplasms
Keywords: Solid tumors, Head and neck non squamous cell carcinoma, breast cancer, PI3K inhibitor, BYL719, paclitaxel
MeSH Terms: conditions — Neoplasms; Breast Neoplasms; Head and Neck Neoplasms | interventions — Alpelisib; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BYL719 and paclitaxel (Experimental): All patients enrolled in the study will receive BYL719 once daily plus weekly paclitaxel
  Interventions: Drug: BYL719; Drug: Paclitaxel

INTERVENTIONS:
Drug: BYL719 — BYL719 will be administered orally once daily on a continuous dosing schedule and dosed on a flat-fixed dose and not adjusted by body weight or body surface area, starting on Day 2 in the dose escalation part and Day 1 in the dose expansion part. In the dose escalation part, the BYL719 starting dose will be 300mg, with anticipated dose escalation to 350mg. In the dose expansion part, BYL719 will be administered at the recommended dose determined in the dose escalation part.
Drug: Paclitaxel — Paclitaxel will be administered once weekly at a dose of 80 mg/m2 i.v. (days 1, 8, 15 and 22) in a 28 day cycle in both dose escalation and expansion.

SUMMARY:
Dose escalation part:to determine the highest dose of BYL719 administered on a daily basis when given in combination with weekly paclitaxel Dose escalation part: to confirm the safety and tolerability of the BYL719 and paclitaxel combination

ELIGIBILITY:
Inclusion criteria For entire trial:

1. - Adult > or = 18 years old
2. - has signed the Informed Consent Form (ICF)
3. - has at least one measurable or non-measurable disease as per RECIST 1.1
4. - has tumor tissue available for the analysis as described in the protocol
5. - has adequate bone marrow and organ function as defined in the protocol
6. - is able to swallow and retain oral medication for the dose escalation part, ALL above PLUS
7. - has a histologically-confirmed, advanced unresectable solid tumors who have progressed on standard therapy (or not been able to tolerate) within three months before screening/baseline visit or for whom no standard anticancer therapy exists.
8. - has an Eastern Cooperative Oncology Group (ECOG) performance status ≤2 For dose expansion part, patient has ALL of above first six criteria PLUS either: 9- has a histologically/cytologically-confirmed HNSCC as detailed in the protocol and an ECOG performance status ≤ 1 or:

   * Patient is a Female with a histologically and/or cytologically confirmed diagnosis of breast cancer as detailed in the protocol and an ECOG performance status ≤ 1

Common exclusion criteria to Dose escalation and Dose expansion parts:

1. - has received previous treatment with a PI3K or AKT inhibitor as described in the protocol
2. - has a known hypersensitivity to paclitaxel or other products containing Cremophor
3. - has a contraindication to use the standard pre-treatment for paclitaxel
4. - has a primary central nervous system (CNS) tumor or CNS tumor involvement as detailed in the protocol
5. - has not recovered to grade 1 or better (except alopecia) from related side effects of any prior antineoplastic therapy
6. - has received radiotherapy > or = 4 weeks prior to starting study drugs, with exception of palliative radiotherapy, who has not recovered from side effects of such therapy to baseline or Grade ≤ 1 and/or from whom ≥ 30% of the bone marrow was irradiated
7. - has peripheral sensory neuropathy with functional impairment (CTC grade 2 neuropathy or higher)
8. - has undergone major surgery ≤ 4 weeks prior to starting study treatment or who has not recovered from side effects of such procedure
9. - has a clinically significant cardiac disease or impaired cardiac function as detailed in the protocol
10. - is currently receiving medication with a known risk of prolonging the QT interval or inducing Torsades de Pointes (TdP) and the treatment cannot either be discontinued or switched to a different medication prior to starting study drug treatment
11. - has diabetes mellitus requiring insulin treatment and/or with clinical signs
12. - has impaired gastrointestinal (GI) function or GI disease as described in the protocol
13. - has a known positive serology for human immunodeficiency virus (HIV), active Hepatitis B, and/or active Hepatitis C infection
14. - has any other condition that would, in the Investigator's judgment, preclude patient's participation in the clinical study due to safety concerns or compliance with clinical study procedures
15. - is currently receiving treatment with drugs known to be moderate or strong inhibitors or inducers of isoenzymes CYP3A or CYP2C8 as detailed in the protocol
16. - is currently receiving treatment with agents that are metabolized solely by CYP3A and/or have a narrow therapeutic window
17. - has a history of another malignancy within 2 years prior to starting study treatment, except cured basal cell carcinoma of the skin or excised carcinoma in situ of the cervix
18. - Patient has a history of non-compliance to medical regimen or inability to grant consent
19. - Pregnant or nursing (lactating) women
20. - does not apply highly effective contraception during the study and through the duration as defined in the protocol

For the HNSCC patient's cohort additional exclusion criteria are:

21- Treatment with more than one prior chemotherapy for recurrent/metastatic disease as detailed in the protocol 22- Prior taxane treatment for metastatic disease additional exclusion criteria for breast cancer patients' cohort:

- has received any prior cytotoxic therapy for the inoperable locally advanced (recurrent or progressive) or metastatic disease, or who had a progression/recurrent disease within 6 months after completion of an adjuvant/neoadjuvant therapy as described in the protocol

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2014-03-05 (Actual); Primary Completion 2016-08-19 (Actual); Study Completion 2016-08-19 (Actual)

PRIMARY OUTCOMES:
Dose escalation : Dose Limiting Toxicity (DLT) | Cycle 1 (28 days)
  A dose-limiting toxicity (DLT) is an adverse event or abnormal laboratory value assessed as being unrelated to disease, disease progression, inter-current illness, or concomitant medications, and that occurs within the first cycle of treatment with BYL719 plus paclitaxel and meets any of the pre-defined criteria.
Dose expansion : Number of patients with adverse events as a measure of safety and tolerability | Screening, every 28 days until 30 days after last dose
  type, intensity, severity and seriousness of adverse events according to the NCI CTC AE v4.03. Dose interruptions, reductions and dose intensity.

SECONDARY OUTCOMES:
Dose escalation:Number of patients with adverse events as a measure of safety and tolerability | Screening, every 28 days until 30 days after last dose
  type, intensity, severity and seriousness of adverse events according to the NCI CTC AE v4.03. Dose interruptions, reductions and dose intensity.
Dose escalation : BYL719 and Paclitaxel Plasma concentrations | Cycle 1 Day 1, Cycle 1 Day 2, Cycle 1 Day 8, Cycle 1 Day 9
  Plasma concentration time profiles of BYL719 and paclitaxel. Plasma PK parameters of paclitaxel (single agent vs. combination) and BYL719 (steady state in combination with paclitaxel).
Dose expansion: Clinical benefit Rate in the breast cancer cohort | Baseline, every 8 weeks (Breast cancer patients) from start of treatment until first documented disease progression up to 2 years
  Clinical benefit rate is defined as the proportion of patients with a best overall response of complete response (CR) or partial response (PR) or stable disease (SD) for more than 24 weeks of duration of response.
Dose expansion: Progression free survival | Baseline, every 6 weeks (head-and-neck squamous cell carcinoma (HNSCC) patients) or every 8 weeks (Breast cancer patients) from start of treatment until first documented disease progression up to 2 years
  Progression-free survival is defined as the time from start date of study treatment until objective tumor progression or death from any cause
Dose expansion: Overall response rate | Baseline, every 6 weeks (HNSCC patients) or every 8 weeks (Breast cancer patients) from start of treatment until first documented disease progression up to 2 years
  Overall response rate is defined as the proportion of patients with a best overall response of complete response (CR) or partial response (PR), based on RECIST 1.1 criteria and the investigator assessment.
Dose expansion : Duration of Response | Baseline, every 6 weeks (HNSCC patients) or every 8 weeks (breast cancer patients) from start of treatment until first documented disease progression up to 2 years
  Duration of response is defined as the time of first occurrence of CR or PR until the date of the first documented disease progression or death due to the disease.
Dose expansion: Plasma pharmacokinetics of BYL719 given in combination with paclitaxel in breast cancer and HNSCC patients | Cycle 1 Day 1, Cycle 1 Day 8, Cycle 2 Day 15, and Day 1 of each subsequent Cycle
  Plasma concentration time profiles of BYL719 and appropriate individual PK parameters.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (5):
- United States (2):
  - Highlands Oncology Group, Fayetteville, Arkansas
  - Horizon Oncology Center BioAdvance, Lafayette, Indiana
- Novartis Investigative Site, Toulouse, France
- Novartis Investigative Site, Milan, MI, Italy
- Novartis Investigative Site, Barcelona, Catalonia, Spain

REFERENCES:
- [Derived] Rodon J, Curigliano G, Delord JP, Harb W, Azaro A, Han Y, Wilke C, Donnet V, Sellami D, Beck T. A Phase Ib, open-label, dose-finding study of alpelisib in combination with paclitaxel in patients with advanced solid tumors. Oncotarget. 2018 Aug 3;9(60):31709-31718. doi: 10.18632/oncotarget.25854. eCollection 2018 Aug 3. PMID 30167089
- See also: Novartis results database — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=16327